CLINICAL TRIAL: NCT02731690
Title: A Phase 2 Open-label Study to Evaluate the Safety of Aceneuramic Acid Extended Release (Ace-ER) Tablets in GNE Myopathy (GNEM) (Also Known as Hereditary Inclusion Body Myopathy (HIBM)) Patients With Severe Ambulatory Impairment
Brief Title: A Study to Evaluate the Safety of Aceneuramic Acid Extended Release (Ace-ER; UX001) Tablets in Glucosamine (UDP-N-acetyl)-2-Epimerase (GNE) Myopathy (GNEM) (Also Known as Hereditary Inclusion Body Myopathy [HIBM]) Patients With Severe Ambulatory Impairment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX001-CL203
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Hereditary Inclusion Body Myopathy; Distal Myopathy With Rimmed Vacuoles; Distal Myopathy, Nonaka Type; GNE Myopathy; Quadriceps Sparing Myopathy; Inclusion Body Myopathy 2
Keywords: GNE Myopathy; Nonaka; GNEM; Hereditary Inclusion Body Myopathy; HIBM; DMRV; QSM
MeSH Terms: conditions — Distal myopathy, Nonaka type

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label UX001, 6g/day (Experimental)
  Interventions: Drug: Aceneuramic Acid Extended-Release

INTERVENTIONS:
Drug: Aceneuramic Acid Extended-Release — oral tablets
  Other Names: Ace-ER; Sialic Acid Extended Release; UX001

SUMMARY:
The primary objective of this Phase 2 study is to evaluate the safety of open-label 6 g/day Ace-ER in GNEM participants with severe ambulatory impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years old
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and before any research-related procedures are conducted
* Have a documented diagnosis of GNEM, HIBM, distal myopathy with rimmed vacuoles (DMRV), or Nonaka disease due to previously demonstrated mutations in the gene encoding the GNE/N-acetylmannosamine kinase (MNK) enzyme (genotyping will not be conducted in this study).
* Should meet the criteria for severe ambulatory impairment defined below:

  * Unable to rise from a seated position to standing without help from another person, assistive device(s), stationary object, or other support AND
  * Unable to walk without the assistance of another person OR if able to walk (use of assistive device(s) permitted), requires at least 2 minutes to walk 40 meters (one full lap of the 6-minute walk test [6MWT] course) AND
  * Use of wheelchair or scooter for activities outside of the home or unable to leave the home independently
* Willing and able to comply with all study procedures
* Participants of child-bearing potential or with partners of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use highly effective method of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation or true abstinence (when this is in line with the preferred and usual lifestyle of the subject) which means not having sex because the subject chooses not to), from the period following the signing of the informed consent through 30 days after last dose of study drug
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause for at least two years, have had tubal ligation at least one year prior to Screening, or who have had a total hysterectomy or bilateral salpingo-oophorectomy

Exclusion Criteria:

* Ingestion of N-acetyl-D-mannosamine (ManNAc), SA, or related metabolites; intravenous immunoglobulin (IVIG); or anything that can be metabolized to produce SA in the body within 60 days prior to the Screening Visit
* Prior participation in a clinical trial involving treatment with Ace-ER/placebo and/or Sialic Acid immediate release (SA-IR) in the past year
* Has had any hypersensitivity to aceneuramic acid or its excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
* Has serum transaminase (i.e. aspartate aminotransferase [AST] or gamma-glutamyl transpeptidase [GGT]) levels greater than 3X the upper limit of normal (ULN) for age/gender, or serum creatinine of greater than 2X ULN at Screening
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or anticipated requirement for any investigational agent prior to completion of all scheduled study assessments
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe participation in the study
* Has a concurrent disease, active suicidal ideation, or other condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or would affect safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- United States (3):
  - University of California, Irvine, Orange, California
  - Washington University, St. Louis, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
- University Alexandrovska, Bulgaria, Sofia, Bulgaria
- McMaster University, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- UX001 6g/Day: Open-label UX001 6000 mg (6 g) total daily dose administered orally divided into a 3-times-daily regimen.
Period: Overall Study
Arm/Group | UX001 6g/Day
Started | 42
Completed | 12
Not Completed | 30
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Discontinuation of Study by Sponsor | 26

BASELINE CHARACTERISTICS:
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  Asian | 2
  Other (Not Specified) | 9
Glucosamine (UDP-N-acetyl)-2-epimerase Myopathy Functional Activities Scale(GNEM-FAS) Mobility Score [Mean (Standard Deviation); unit: units on a scale] — GNEM-FAS Expanded Version Mobility subscale scores have 13 items and range from 0 to 52 with higher scores representing greater mobility. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  units on a scale
    number analyzed (Participants) | 41
    (all) | 10.63 (7.816)
GNEM-FAS Upper Extremity Domain Score [Mean (Standard Deviation); unit: units on a scale] — GNEM-FAS Expanded Version Upper Extremity subscale scores have 9 items and range from 0 to 36 with higher scores representing more skilled, independent use of the arms during functional activity performance. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  units on a scale
    number analyzed (Participants) | 41
    (all) | 15.20 (8.897)
GNEM-FAS Self-Care Domain Score [Mean (Standard Deviation); unit: units on a scale] — GNEM-FAS Expanded Version Self-Care subscale scores have 8 items range from 0 to 32 with higher scores representing greater independence with functional care activities. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  units on a scale
    number analyzed (Participants) | 41
    (all) | 13.00 (7.413)
GNEM-FAS Total Score [Mean (Standard Deviation); unit: units on a scale] — GNEM-FAS Expanded Version Total Score were calculated as the sum of the subscale Scores range from 0 to 120 with higher scores representing greater independence with functional activities. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  units on a scale
    number analyzed (Participants) | 41
    (all) | 38.83 (23.116)
Hand-Held Dynamometry (HHD) Raw Strength: Average Grip [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kilogram-force [kgf]) for each was recorded. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  kgf
    number analyzed (Participants) | 41
    (all) | 5.535 (7.6778)
HHD Raw Strength: Average Shoulder Abduction [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  kgf
    number analyzed (Participants) | 41
    (all) | 3.880 (4.4583)
HHD Raw Strength: Average Wrist Extension [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  kgf
    number analyzed (Participants) | 41
    (all) | 3.532 (3.5177)
HHD Lower Extremity Muscle Strength: Average Knee Extension [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  kgf
    number analyzed (Participants) | 41
    (all) | 10.50 (8.001)
HHD Raw Strength: Key Pinch [Mean (Standard Deviation); unit: kgf] — Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
  kgf
    number analyzed (Participants) | 41
    (all) | 1.790 (2.1614)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Discontinuation
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug, whether or not considered drug related. An SAE or serious suspected adverse reaction is an AE or suspected adverse reaction that at any dose, in the view of either the Investigator or Ultragenyx, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect. TEAEs were defined as any AE that occurred after the first dose of study drug.
Time Frame: 48 Weeks (plus 30 [+5] days for participants not enrolling in extension study)
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
Participants
  TEAEs | 30
  Serious TEAEs | 1
  TEAEs Causing Study Drug Discontinuation | 1
  TEAEs Causing Study Discontinuation | 1

2. Secondary Outcome: Number of Participants Taking Prior and Concomitant Medications
Description: Prior medications are any medications which started before the date of the first dose of investigational product. Concomitant medications are any medications that are taken on or after the date of the first dose of investigational product excluding concomitant medications started after the date of the last dose of investigational product.
Time Frame: 48 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
Participants
  Prior Medications | 31
  Concomitant Medications | 33

3. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline In Physical Examinations
Description: Complete physical examinations included assessments of general appearance; head, eyes, ears, nose, and throat; the cardiovascular, dermatologic, lymphatic, respiratory, GI, musculoskeletal, and neurologic systems. The neurologic system examination included assessments of cognition, cranial nerves, motor function, coordination and gait, reflexes, and sensory function. Brief physical examinations included assessments of general appearance, cardiovascular and respiratory systems, and a focus on any presenting complaints.
Time Frame: 48 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
participants | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline In Vital Signs
Description: Vital signs included seated systolic blood pressure and diastolic blood pressure, heart rate, respiration rate, and temperature.
Time Frame: 48 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
participants | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline In Clinical Laboratory Results
Description: The clinical laboratory evaluations performed included serum chemistry, complete blood count (hematology), and urinalysis.
Time Frame: 48 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
participants
  Hematology | 0
  Clinical Chemistry | 2
  Urinalysis | 0

6. Secondary Outcome: Number of Participants With Overall Suicidal Behaviors and/or Ideation at Baseline and Post-Baseline
Description: As evaluated by the Columbia Suicide Severity Rating Scale (C-SSRS), a participant-rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses).
Time Frame: 48 weeks
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 42
Participants
  Overall Suicidal Behaviors: Baseline | 1
  Overall Suicidal Behaviors: Post-Baseline | 0
  Non-Suicide Self-Injurious Behavior: Baseline | 0
  Non-Suicide Self-Injurious Behavior: Post-Baseline | 0
  Completed Suicide: Post-Baseline | 0
  Overall Suicidal Ideation: Baseline | 7
  Overall Suicidal Ideation: Post-Baseline | 1

7. Secondary Outcome: Change From Baseline in GNEM-FAS Expanded Version Mobility Domain Subscale Scores Over Time
Description: GNEM-FAS Expanded Version Mobility subscale scores have 13 items and range from 0 to 52 with higher scores representing greater mobility. Analyzed using a repeated measure generalized estimation equation (GEE) model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
units on a scale
  Week 12 | 0.16 [-0.33 to 0.64]
  Week 24 | -0.65 [-1.56 to 0.27]
  Week 36 | -0.69 [-1.57 to 0.18]
  Week 48 | -1.03 [-2.15 to 0.09]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.5303, GEE model — Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.1646, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.1189, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.0706, GEE model — [p-value comment as in outcome 7, analysis 1]

8. Secondary Outcome: Change From Baseline in GNEM-FAS Expanded Version Upper Extremity Domain Subscale Scores Over Time
Description: GNEM-FAS Expanded Version Upper Extremity subscale scores have 9 items and range from 0 to 36 with higher scores representing more skilled, independent use of the arms during functional activity performance. Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
units on a scale
  Week 12 | 0.57 [-0.05 to 1.19]
  Week 24 | -0.62 [-1.50 to 0.26]
  Week 36 | -0.51 [-1.58 to 0.55]
  Week 48 | -1.91 [-3.93 to 0.11]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.0715, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.1697, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.3428, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.0642, GEE model — [p-value comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in GNEM-FAS Expanded Version Self-Care Domain Subscale Scores Over Time
Description: GNEM-FAS Expanded Version Self-Care subscale scores have 8 items range from 0 to 32 with higher scores representing greater independence with functional care activities. Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
units on a scale
  Week 12 | -0.39 [-0.79 to 0.01]
  Week 24 | -0.71 [-1.43 to 0.01]
  Week 36 | -0.83 [-1.64 to -0.02]
  Week 48 | -0.40 [-1.78 to 0.98]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.0568, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.0533, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.0459, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.5678, GEE model — [p-value comment as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in GNEM-FAS Expanded Version Total Scores Over Time
Description: GNEM-FAS Expanded Version Total Score were calculated as the sum of the subscale Scores range from 0 to 120 with higher scores representing greater independence with functional activities. Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
units on a scale
  Week 12 | 0.35 [-0.89 to 1.58]
  Week 24 | -1.95 [-3.87 to -0.03]
  Week 36 | -2.02 [-4.46 to 0.42]
  Week 48 | -3.34 [-6.90 to 0.22]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.5810, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.0465, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.1047, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.0661, GEE model — [p-value comment as in outcome 7, analysis 1]

11. Secondary Outcome: Change From Baseline in HHD Raw Strength (Grip) Over Time
Description: Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded. Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
kgf
  Week 12 | 0.258 [-0.103 to 0.620]
  Week 24 | 0.128 [-0.377 to 0.632]
  Week 36 | 0.038 [-0.724 to 0.799]
  Week 48 | -0.261 [-1.325 to 0.803]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.1615, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.6201, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.9229, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.6307, GEE model — [p-value comment as in outcome 7, analysis 1]

12. Secondary Outcome: Change From Baseline in HHD Raw Strength (Shoulder Abductors) Over Time
Description: as for outcome 11
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
kgf
  Week 12 | 0.339 [0.085 to 0.592]
  Week 24 | 0.379 [-0.228 to 0.987]
  Week 36 | 0.437 [0.075 to 0.800]
  Week 48 | -0.277 [-0.698 to 0.144]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.0088, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.2213, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.0180, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.1970, GEE model — [p-value comment as in outcome 7, analysis 1]

13. Secondary Outcome: Change From Baseline in HHD Raw Strength (Wrist Extensors) Over Time
Description: as for outcome 11
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
kgf
  Week 12 | 0.235 [-0.024 to 0.495]
  Week 24 | 0.152 [-0.486 to 0.791]
  Week 36 | 0.358 [-0.228 to 0.943]
  Week 48 | -0.123 [-0.924 to 0.678]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.0752, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority — Analyzed using a repeated measure GEE model, which includes the change from baseline as the dependent variable, visit as a fixed factor, and the baseline value as a covariate. Compound symmetry is used as the covariance structure; p = 0.6403, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority — [test comment as in outcome 13, analysis 2]; p = 0.2316, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.7635, GEE model — [p-value comment as in outcome 7, analysis 1]

14. Secondary Outcome: Change From Baseline in HHD Muscle Strength in Knee Extensors Over Time
Description: as for outcome 11
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kgf
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
kgf
  Week 12 | 0.80 [-0.12 to 1.73]
  Week 24 | 1.35 [0.36 to 2.33]
  Week 36 | 2.05 [0.52 to 3.58]
  Week 48 | 2.45 [0.01 to 4.88]
Statistical Analysis 1: Comparison: UX001 6g/Day; Week 12; Test type: Superiority; p = 0.0872, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: UX001 6g/Day; Week 24; Test type: Superiority; p = 0.0073, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: UX001 6g/Day; Week 36; Test type: Superiority; p = 0.0086, GEE model — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 4: Comparison: UX001 6g/Day; Week 48; Test type: Superiority; p = 0.0489, GEE model — [p-value comment as in outcome 7, analysis 1]

15. Secondary Outcome: Change From Baseline in HHD Raw Strength (Key Pinch) Over Time
Description: Hand held dynamometry testing was used to measure strength. The maximum voluntary isometric contraction against a dynamometer was used to measure bilateral strength in the following muscle groups: shoulder abductors, wrist extensors and knee extensors. Specialized dynamometers for the measurement of grip and key pinch strength were also used. The total force (in kgf) for each was recorded.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Full Analysis Set: all participants with a baseline measurement and at least 1 postbaseline measurement at given time point.
Measure: Mean (Standard Deviation); unit: kgf
Arm/Group | UX001 6g/Day
Number analyzed (Participants) | 41
kgf
  Week 12 | 0.110 (0.7083)
  Week 24: number analyzed (Participants) | 30
  Week 24 | 0.112 (0.6534)
  Week 36: number analyzed (Participants) | 23
  Week 36 | 0.049 (0.8090)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 0.318 (0.9509)

ADVERSE EVENTS:
Time Frame: 48 Weeks (plus 30 [+5] days for participants not enrolling in extension study)
Groups:
- Ace-ER 6 g/Day: Open-label UX001 6000 mg (6 g) total daily dose administered orally divided into a 3-times-daily regimen.
Arm/Group | Ace-ER 6 g/Day
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 26/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=42)
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ace-ER 6 g/Day (N=42)
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT02731690/SAP_000.pdf
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02731690/Prot_001.pdf